CLINICAL TRIAL: NCT00667550
Title: Lower Urinary Tract and Sexual Function in Women Following Surgery for Colorectal Disorders
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Karen Noblett, Associate Professor, University of California, Irvine Medical Center
Other Study IDs: 2007-5995
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2010-07

CONDITIONS: Lower Urinary Tract Symptoms; Colorectal Disorders
Keywords: Lower urinary tract symptoms; Colorectal disorders; Urinary incontinence; Fecal incontinence; Voiding dysfunction; Urgency frequency; Sexual dysfunction; Colorectal malignancies; Inflammatory bowel disease
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Incontinence; Fecal Incontinence; Sexual Dysfunction, Physiological; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prevalence study evaluating lower urinary tract, prolapse, bowel, and sexual symptoms in women with a colorectal disorder who are planning to undergo surgery.

The purpose of this study is to identify the number of women who complain of lower urinary tract and bowel problems, including frequency, urgency, urinary incontinence, fecal incontinence, pain with intercourse, and other sexual problems prior to undergoing surgical management for a colorectal disorder.

DETAILED DESCRIPTION:
Lower urinary tract symptoms, including urinary incontinence, voiding dysfunction, urgency, frequency, fecal incontinence, as well as sexual dysfunction, are directly affected by surgery for colorectal disorders. Increased risk of injury to the urinary tract is a recognized complication of pelvic surgery. These risks are related to the radical nature of pelvic surgery used to treat certain colorectal disorders, including colorectal malignancies and inflammatory bowel disease.

Few studies have looked at the incidence of lower urinary tract symptoms and sexual dysfunction in patients with colorectal conditions before and after surgery.

The primary goal of this study is to determine the prevalence of lower urinary tract symptoms in women undergoing surgery for colorectal ocnditions. We also want to describe the prevalence of these symptoms in different colorectal disorders, and how pelvic surgery impacts these symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with a diagnosis of a colorectal disorder, including rectal prolapse, inflammatory bowel disease such as Crohn's disease, Ulcerative Colitis, and colorectal malignancies planning to undergo surgery
* Females have English as a primary language

Exclusion Criteria:

* Subjects less than 18 years of age
* Subjects unable to give informed consent or complete the validated questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with a diagnosis of a colorectal disorder requiring surgery. Patients must be able to complete the questionnaires in English as the questionnaires are only available and valid in English.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Noblett, M.D., Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States